CLINICAL TRIAL: NCT05289726
Title: Randomized Controlled Clinical Trials to Evaluate the Preventive Effect of Traditional Chinese Medicine TDX105 on Anti-tumor Target Therapy Regorafenib Induced Dermatologic Toxicities
Brief Title: Study on the Prevention of Dermal Toxicity Caused by Regorafenib by Traditional Chinese Medicine TDX105
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: APL21100510010105003002
Record Dates: First submitted 2021-12-10; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Hand and Foot Skin Reaction; Colorectal Cancer Stage IV
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional chinese medicine TDX105 (Experimental): * Experimental group Traditional chinese medicine TDX105 (Dissolve in warm water and then dilute to 600ml and soak hands and feet for 30 minutes each time, once in the morning and evening every day, until the end of the first 8 weeks of treatment with regorafenib)
  * Basic care was the same in both groups, including routine care such as topical use of urea ointment
  Interventions: Drug: Traditional chinese medicine TDX105
- placebo (Placebo Comparator): The control group received placebo granules mixed with dextrin and food coloring (Dissolve in warm water and then dilute to 600ml and soak hands and feet for 30 minutes each time, once in the morning and evening every day, until the end of the first 8 weeks of treatment with regorafenib)
  - Basic care was the same in both groups, including routine care such as topical use of urea ointment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Traditional chinese medicine TDX105 — Experimental group Traditional chinese medicine TDX105
  Arms: Traditional chinese medicine TDX105
Drug: Placebo — he control group received placebo granules mixed with dextrin and food coloring
  Arms: placebo

SUMMARY:
this is an preventive study to evaluate the preventive effect of traditional chinese medicine TDX105 on Regorafenib induced Dermatologic Toxicities

DETAILED DESCRIPTION:
this is an double blinded controlled preventive study to evaluate the preventive effect of this is an preventive traditional chinese medicine TDX105 plus Urea Ointment compared with placebo plus Urea Ointment on Regorafenib induced Dermatologic Toxicities

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed colorectal cancer patients;
2. It is planned to use the targeted drug regorafenib for the first time, and the initial dose is 120mg/d;
3. Performance Status score ≤3;
4. Age ≥18; 5, no intellectual and mental disorders, normal language expression ability, ability to judge their own symptoms

6. Understand and agree to accept the treatment, and sign the informed consent.

Exclusion Criteria:

1. Patients with skin reactions affected by simultaneous use of other targeted drugs (sorafenib, sunitinib, fruquintinib, etc.), chemotherapy drugs (capecitabine, doxorubicin, etc.) or hand-foot radiotherapy;
2. Patients with skin diseases such as eczema, psoriasis and tinea pedis at observed skin sites (namely hands and feet); Patients with skin allergic diseases;
3. Patients in the study who cannot cooperate with the continuation of this treatment;
4. Sudden changes in the patient's condition affected and interfered with the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-04-18 (Estimated); Primary Completion 2022-07-18 (Estimated); Study Completion 2023-04-18 (Estimated)

PRIMARY OUTCOMES:
incidence of grade 3 hand-foot skin reaction | Once a week from the beginning to 2 months
  Evaluation criteria for common adverse events (CTCAE) 5.0

SECONDARY OUTCOMES:
Grade 1-2 hand and foot skin reaction rate | Once a week from the beginning to 2 months
  Evaluation criteria for common adverse events (CTCAE) 5.0
Withdrawal rate of regorafenib within 2 cycles | Once a week from the beginning to 2 months
  Weekly telephone follow-up
progression-free survival | Measures were taken every 2 months from date of randomization until the date of first documented progression, assessed up to 36 months.
  Response Evaluation Criteria In Solid Tumors 1.1
tumor control rate | Measures were taken every 2 months from date of randomization until the date of first documented progression, assessed up to 36 months.
  Response Evaluation Criteria In Solid Tumors 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Chinese academy of Medical sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Do not participate in data sharing

REFERENCES:
- [Derived] Yu S, Hu X, Tan Y, Wang C, Shao Z, Xiao Y, Liu H, Lv J, Li S, Jiang X, Zeng L, Tian A. Prophylactic effect of the traditional Chinese medicine formula danxiong granules (TDX105) on hand-foot skin reaction associated with the antitumor targeted drug regorafenib: a randomized, double-blind, placebo-controlled trial. Front Pharmacol. 2025 Nov 6;16:1641477. doi: 10.3389/fphar.2025.1641477. eCollection 2025. PMID 41282614